CLINICAL TRIAL: NCT02698098
Title: Comparing Health & Social Outcomes Between Opioid-Dependent Individuals in Compulsory Drug Rehabilitation Centers and Voluntary Drug Treatment Clinics in Klang Valley, Malaysia
Brief Title: Comparative Evaluation of PUSPENs and C&Cs
Acronym: PSVCC
Status: Terminated | Type: Observational
Why Stopped: 1) Policy change affecting C&Cs; 2) interm analysis revealing overt differences
Sponsor: University of Malaya (Other)
Collaborators: Yale University (Other); World Bank (Other); Doris Duke Charitable Foundation (Other); National Institute of Mental Health (NIMH) (NIH); The University of New South Wales (Other); Burnet Institute (Other); University of Florida (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1206010403; F30MH105153 (NIH); K24DA017072 (NIH); R01DA025943 (NIH); HIRGA E000001-20001 (Other: Malaysian Ministry of Education (High Impact Research Grant))
Record Dates: First submitted 2016-02-16; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Opioid-Related Disorders
Keywords: Malaysia; Asia; Southeast Asia; Compulsory Drug Detention Centers; Compulsory Centers for Drug Users; Methadone; Drug Relapse; Drug and Narcotic Control; Opiate Substitution Treatment; Prisons
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Compulsory Drug Detention Center: Conventional drug treatment in Malaysia and Southeast Asia including detention for an average of 2 years, including educational and job skills programs and physical education. Medical therapies for treating substance use disorders, such as opioid-agonist treatment (OAT), are unavailable.
- Voluntary Treatment Center: Voluntary drug treatment facilities, called 'Cure and Care' centers in Malaysia, that provide methadone maintenance therapy in addition to psychosocial interventions, recreational programming, and vocational training, among other activities.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone
  Groups: Voluntary Treatment Center

SUMMARY:
This observational study compares the health and social outcomes between opioid-dependent individuals who are either recently released from a compulsory drug detention center (CDDC) or recently discharged from a voluntary treatment center (VTC) providing methadone maintenance therapy, in Malaysia.

DETAILED DESCRIPTION:
In July 2010, the National Anti-Drug Agency of Malaysia (NADA) introduced a non-punitive system of treatment and care for people who use drugs, voluntary treatment centers (VTCs), called 'Cure & Care' clinics, offering free methadone maintenance therapy (MMT) to opioid-dependent drug users. These centers were opened alongside existing compulsory drug detention centers (CDDCs), where people who use drugs continue to be detained involuntarily without access to evidence-based treatment. Given that both of these programs are operated by NADA but espouse vastly different responses to drug use, we compared health and social outcomes between opioid-dependent individuals recently released from CDDCs and recently initiated into MMT in the new VTCs.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual-IV criteria for opioid dependence
* Physically and psychologically capable of understanding and undergoing informed consent process
* Within 90 days of release or discharge and intending to return to Klang Valley region
* For VTC arm, came to the C&C to start MMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted among opioid-dependent individuals initiating MMT in C&C Centers and opioid-dependent individuals being released from Pusat Serenti who consent to participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of opioid use (urine-toxicology) | Year following release from CDDC or discharge from VTC

SECONDARY OUTCOMES:
Occurrence of any drug use (urine-toxicology) | Year following release from CDDC or discharge from VTC
  Includes opioid, amphetamine and benzodiazepine use
Occurrence of amphetamine use (urine-toxicology) | Year following release from CDDC or discharge from VTC
Occurrence of benzodiazepine use (urine-toxicology) | Year following release from CDDC or discharge from VTC
Occurrence of methadone use (urine-toxicology) | Year following release from CDDC or discharge from VTC
  This is a proxy for linkage to methadone therapy
Occurrence of buprenorphine use (urine-toxicology) | Year following release from CDDC or discharge from VTC
  This is a proxy for linkage to buprenorphine therapy
Occurrence of no-methadone use (urine-toxicology) | Year following release from CDDC or discharge from VTC
  This is a proxy for retention in methadone therapy

OTHER OUTCOMES:
Occurrence of drug or methadone use (self-report) | Year following release from CDDC or discharge from VTC
  Sub-measures include opioid use, any drug use (opioid, amphetamine, benzodiazepine), methadone use, buprenorphine use
Addiction Severity (self-report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Occurrence of non-fatal overdose (self-report) | Year following release from CDDC or discharge from VTC
Rates of injection-related HIV risk behaviors (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Rates of sex-related HIV risk behaviors (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Opioid cravings (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Motivation to change drug use (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Police harassment (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Health-related quality of life (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Social Support (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Occurrence of HIV seroconversion (antibody test) | Year following release from CDDC or discharge from VTC
Rates of employment (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Total monthly income (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Days of criminal activity (self report) | Compared at 3, 6, 9 and 12-months following release from CDDC or discharge from VTC
Detention in CDDC/Incarceration in jail or prison | Year following release from CDDC or discharge from VTC

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, MD, Principal Investigator — Yale University; Adeeba Kamarulzaman, FRACP, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: Yes
See links at end of this record for accessing de-identified data and documentation.

REFERENCES:
- [Derived] Wegman MP, Altice FL, Kaur S, Rajandaran V, Osornprasop S, Wilson D, Wilson DP, Kamarulzaman A. Relapse to opioid use in opioid-dependent individuals released from compulsory drug detention centres compared with those from voluntary methadone treatment centres in Malaysia: a two-arm, prospective observational study. Lancet Glob Health. 2017 Feb;5(2):e198-e207. doi: 10.1016/S2214-109X(16)30303-5. Epub 2016 Dec 8. PMID 27964869
- See also: Link to dataverse site with protocol, study questionnaires, individual de-identified data and analytic code — http://dx.doi.org/10.7910/DVN/RO34OK
- Available data/document: Study Protocol — http://dx.doi.org/10.7910/DVN/RO34OK
- Available data/document: Individual Participant Data Set — http://dx.doi.org/10.7910/DVN/RO34OK
- Available data/document: Analytic Code — http://dx.doi.org/10.7910/DVN/RO34OK